CLINICAL TRIAL: NCT03857867
Title: A Prospective, Randomized, Staggered-onset, Double Blinded, Sham-Controlled Study to Evaluate Peripheral Vibrotactile Coordinated Reset (CR) Stimulation for Parkinson's Disease
Brief Title: Evaluation of Using Vibrotactile Coordinated Reset for Management of Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid 19
Sponsor: Peter Tass, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Peter Tass, MD, PhD, Professor of Neurosurgery, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-47775
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Tactile Stimulation Glove (Experimental): Patient will receive active stimulation for a minimum of 3 months and a maximum of 13 months
  Interventions: Device: Tactile Stimulation Glove

INTERVENTIONS:
Device: Tactile Stimulation Glove — A glove device produces non-painful sensory (tactile) vibratory stimulation to the fingertips of Parkinson's patients.

SUMMARY:
This is a study to evaluate peripheral vibrotactile coordinated reset stimulation for Parkinson's disease seeks to explore the safety and efficacy of an experimental non-invasive method to aid in the symptoms of Parkinson's disease. The purpose of the study is to verify the safety and tolerability of non-painful sensory (tactile) vibratory stimulation delivered to the fingertips of patients with Parkinson's disease.

DETAILED DESCRIPTION:
This study aims to evaluate the safety and efficacy of a non-invasive, experimental method to aid in the symptoms of Parkinson's disease. A glove device produces non-painful sensory (tactile) vibratory stimulation to the fingertips of Parkinson's patients. Vibrotactile coordinated reset (vCR) will help investigators compare durability and efficacy of the tactile stimulation to current medical therapy. Participants will receive vCR for a minimum of 3 months and a maximum of 13 and motor ability will be recorded. If the results of this study suggest that vibrotactile CR stimulation is safe and effective for the treatment of Parkinson's disease, this non-invasive treatment approach would have a substantial impact on Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Diagnosis of idiopathic Parkinson's disease.
3. Levodopa responsiveness as defined by at least a 30% reduction in Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) motor subscale (excluding tremor scores) in the ON vs off medication state.
4. Willing to participate in the vibrotactile stimulation sessions for 2 consecutive days initially and willing to return for follow-up visits
5. Able to provide informed consent.
6. Appropriate social support

Exclusion Criteria:

1. Hoehn and Yahr stage greater than 3 in the on medication state
2. Presence of other forms of non-idiopathic parkinsonism, including but not limited to atypical parkinsonism, medication induced parkinsonism, vascular Parkinsonism
3. Any illness that in the investigator's opinion precludes participation in the study
4. Subjects unable to communicate with the investigator and staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pfeifer KJ, Kromer JA, Cook AJ, Hornbeck T, Lim EA, Mortimer BJP, Fogarty AS, Han SS, Dhall R, Halpern CH, Tass PA. Coordinated Reset Vibrotactile Stimulation Induces Sustained Cumulative Benefits in Parkinson's Disease. Front Physiol. 2021 Apr 6;12:624317. doi: 10.3389/fphys.2021.624317. eCollection 2021. PMID 33889086

RESULTS

PARTICIPANT FLOW:
Groups:
- Tactile Stimulation Glove: Patient receive Tactile Stimulation Glove stimulation for a minimum of 3 months and a maximum of 13 months. The glove device produces non-painful sensory (tactile) vibratory stimulation to the fingertips of Parkinson's patients.
Period: Overall Study
Arm/Group | Tactile Stimulation Glove
Started | 7
Completed | 6
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol are included in the analysis.
Groups:
- Tactile Stimulation Glove: Patient receive Tactile Stimulation Glove stimulation for a minimum of 3 months and a maximum of 13 months.
Arm/Group | Tactile Stimulation Glove
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.33 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
MDS-UPDRS Baseline [Mean (Standard Deviation); unit: units on a scale] — The MDS-UPDRS III is the sum of 33 scores that evaluate Parkinson's disease motor symptoms on a scale from 0 to 4 points. A score of 0 indicated no symptom is present and a maximum score of 4 indicates the most severe symptom, the total scale range is 0-132, where higher scores indicate more severe symptoms.
  units on a scale | 38.33 (5.93)
Levodopa equivalent daily dose (LEDD) [Mean (Standard Deviation); unit: mg/day] — LEDD is calculated as a sum of each Parkinson's medication in mg a day
  mg/day | 711.50 (207.85)
Electroencephalography (EEG) sensorimotor relative power activity [Mean (Standard Deviation); unit: percentage of total power] — Baseline EEG was recorded. EEG source estimation was computed using Standardized low-resolution brain electromagnetic tomography analysis (sLORETA) and was restricted to the sensorimotor region. Power spectral density (PSD) was calculated for each frequency band (Delta: 2-4 Hz; Theta: 5-7 Hz; Alpha: 8-12 Hz; Low Beta: 13-16 Hz; Mid Beta: 17-20 Hz; High Beta: 21-30 Hz; Gamma: 31-50 Hz). Relative power (RP) was calculated by taking the sum of each frequency and dividing it by the total power (2-50 Hz) expressed as a percentage. High beta power was the frequency band of interest for analysis. Population: 5 out of 6 participants EEG were able to be analyzed. One patients EEG was not recorded due to covid-19
  percentage of total power
    number analyzed (Participants) | 5
    (all) | 0.079 (0.036)

OUTCOME MEASURES:

1. Primary Outcome: Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III Score
Description: The MDS-UPDRS III is the sum of 33 scores that evaluate Parkinson's disease motor symptoms on a scale from 0 to 4 points. A score of 0 indicated no symptom is present and a maximum score of 4 indicates the most severe symptom, the total scale range is 0-132, where higher scores indicate more severe symptoms.
Time Frame: Baseline, 3 months
Population: Participants who completed baseline and the 3 month follow up are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Tactile Stimulation Glove: Patients receive Tactile Stimulation for 3 months
Arm/Group | Tactile Stimulation Glove
Number analyzed (Participants) | 6
score on a scale
  Baseline | 38.33 (5.93)
  3 months | 32.33 (7.80)

2. Secondary Outcome: Levodopa Equivalent Daily Dose
Description: Levodopa equivalent daily dose (LEDD) was measured at baseline and after 3 months of vibrotactile coordinated reset therapy. LEDD is calculated as a sum of each Parkinson's medication.
Time Frame: Baseline, 3 months
Population: Participants who completed baseline and the 3 month protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Tactile Stimulation Glove
Number analyzed (Participants) | 6
mg/day
  Baseline LEDD | 711.50 (207.85)
  3 month LEDD | 644.83 (229.85)

3. Secondary Outcome: Electroencephalography (EEG) Sensorimotor Relative Power Activity
Description: Measure Description: Baseline EEG was recorded. EEG source estimation was computed using Standardized low-resolution brain electromagnetic tomography analysis (sLORETA) and was restricted to the sensorimotor region. Power spectral density (PSD) was calculated for each frequency band (Delta: 2-4 Hz; Theta: 5-7 Hz; Alpha: 8-12 Hz; Low Beta: 13-16 Hz; Mid Beta: 17-20 Hz; High Beta: 21-30 Hz; Gamma: 31-50 Hz). Relative power (RP) was calculated by taking the sum of each frequency and dividing it by the total power (2-50 Hz) expressed as a percentage. High beta power was the frequency band of interest for analysis.
Time Frame: Baseline, 3 months
Population: Participants who completed the baseline and 3 month EEG were included in the analysis
Measure: Mean (Standard Deviation); unit: percentage of total power
Arm/Group | Tactile Stimulation Glove
Number analyzed (Participants) | 5
percentage of total power
  Baseline high beta relative power | 0.079 (0.036)
  3 months high beta relative power | 0.058 (0.025)

ADVERSE EVENTS:
Time Frame: Up to 13 months
Arm/Group | Tactile Stimulation Glove
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
The study did not meet its accrual goal of 20 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT03857867/Prot_SAP_000.pdf